CLINICAL TRIAL: NCT00412022
Title: Phase III Randomized Study of the Effects on Bone Mineral Density of Tamoxifen, Letrozole, and Letrozole + Zoledronic Acid as Adjuvant Treatment of Patients With Early Breast Cancer; VERSION 2 AMENDED Phase 3 Study of Triptorelin and Tamoxifen, Letrozole, or Letrozole + Zoledronic Acid in Adjuvant Treatment of Premenopausal Endocrine Responsive Breast Cancer Patients.
Brief Title: HOBOE: A Phase 3 Study of Adjuvant Triptorelin and Tamoxifen, Letrozole, or Letrozole and Zoledronic Acid in Premenopausal Patients With Breast Cancer.
Acronym: HOBOE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Cancer Institute, Naples (Other)
Collaborators: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HOBOE
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer
Keywords: early breast cancer; adjuvant therapy; premenopause; premenopausal; menopausal status; postmenopause; bone mineral density; hormone sensitive; aromatase inhibitors; letrozole; disease-free survival
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Triptorelin Pamoate; Letrozole; Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Active Comparator): Triptorelin 3.75 mg IM every 4 weeks and Tamoxifen 20 mg daily, for 5 years
  Interventions: Drug: tamoxifen; Drug: triptorelin
- B (Active Comparator): Triptorelin 3.75 mg IM every 4 weeks and Letrozole 2.5 mg daily, for 5 years
  Interventions: Drug: triptorelin; Drug: letrozole
- C (Experimental): Triptorelin 3.75 mg IM every 4 weeks and Letrozole 2.5 mg daily for 5 years + zoledronic acid 4 mg every 6 months.
  Interventions: Drug: triptorelin; Drug: letrozole; Drug: zoledronic acid

INTERVENTIONS:
Drug: tamoxifen — 20 mg daily for 5 years
  Arms: A
Drug: triptorelin — Premenopausal patients will receive triptorelin 3.75 mg IM at the beginning of therapy and every 4 weeks for 5 years or up to age 55
Drug: letrozole — 2.5 mg daily for 5 years
  Arms: B; C
Drug: zoledronic acid — 4 mg every 6 months
  Arms: C

SUMMARY:
The HOBOE study was amended in November 2009, and, after reaching enrollment of the first 500 patients, the study began recruiting premenopausal patients only. The primary objective of the extended study is to compare disease free survival in premenopausal patients with early breast cancer. Patients receive triptorelin and are randomized in a 1:1:1 fashion to receive tamoxifen or letrozole, or letrozole + zoledronic acid.

The purpose of the HOBOE study, Version 1, was to compare the adjuvant hormonal therapy treatments of Tamoxifen, Letrozole and Letrozole + Zoledronate for their effects on bone loss in breast cancer patients. Postmenopausal and premenopausal patients were eligible, the latter also receiving monthly triptorelin. Upon reaching the enrollment of the first 500 patients in March 2010, the study began recruiting premenopausal patients only.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of breast cancer
* Surgical resection of breast cancer (breast conserving surgery or mastectomy)
* No evidence of disease
* Indication for adjuvant hormonal therapy (ER and/or PgR positive with IHC exam in at least 1% of primary tumor cells, according to St. Gallen criteria)
* Patient age at least 18 years
* Written informed consent . Premenopausal status defined as LMP within 12 months of randomization (FSH, LH will not be considered as determinants of menopausal status due the chemotherapy induced reversible ovarian suppression)

Please note that patients who have received neoadjuvant or adjuvant chemotherapy and/or locoregional radiation therapy may be included in the study

Exclusion Criteria:

* Performance status (ECOG)>2.
* Previous or concomitant malignancy (with the exception of adequately treated nonmalignant skin cancer and carcinoma in situ of the uterine cervix
* Metastatic breast cancer
* Creatinine > 1.25 times the value of upper normal limit
* Pregnant or lactating females
* Clinical or radiologic evidence of bone fractures
* Treatment with systemic cortisone therapy within 12 months prior to randomization
* Treatment with drugs that could alter bone metabolism (calcitonin, mithramycin, gallium nitrate) within 2 weeks prior to randomization
* Previous treatment with tamoxifen or aromatase inhibitors
* AST and/or ALT > 3 times the value of upper normal limit with clinical and laboratory findings that indicate a grade of hepatic insufficiency that could potentially increase the risk of assuming letrozole
* Any concomitant conditions that would, in the Investigator's opinion, contraindicate the use of any of the drugs used in this study
* Inability to provide informed consent
* Inability to comply with followup
* Patient undergoing invasive dental work at time of baseline evaluation or foreseen during the course of adjuvant therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1294 (Actual)
Dates: Start 2004-03; Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
disease free survival in premenopausal patients | observation period is 10 years from initiation of treatment
bone mineral density | 12 months from initiation of therapy

SECONDARY OUTCOMES:
Bone mineral density measured | yearly after first year of therapy
disease free survival in postmenopausal patients | observation period is 10 years from initiation of treatment
overall survival | observation period is 10 years from initiation of treatment
toxicity of letrozole + triptorelin and letrozole + zoledronic acid + triptorelin in premenopausal patients | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Andrea De Matteis, M.D., Principal Investigator — NCI Naples, Division of Medical Oncology C; Ciro Gallo, M.D., Ph.D., Principal Investigator — University of Campania Luigi Vanvitelli; Francesco Perrone, M.D., Ph.D., Principal Investigator — NCI Naples, Clinical Trials Unit
Locations (20):
- Italy (20):
  - S. Giuseppe Moscati, Avellino, AV
  - Azienda Ospedaliera Treviglio - Caravaggio, Treviglio, BG
  - Azienda Ospedaliera G. Rummo, Benevento, BN
  - Ospedale Senatore Antonio Perrino, Brindisi, BR
  - Istituto Romagnolo per lo Studio e la Cura dei Tumori, Meldola, FC
  - Presidio Ospedaliero Di Saronno Aziendo Ospedaliera di Busto Arsizio, Saronno, VA
  - Ospedale Santa Maria Annunziata, Bagno a Ripoli
  - Istituto Nazionale per la ricerca Sul Cancro, Genova
  - Ospedale Riuniti, Livorno
  - Ospedale Unico della Versilia, Lucca
  - Istituto Nazionale dei Tumori,, Napoli
  - Ospedale Cardarelli, Napoli
  - Seconda Università di Napoli, Napoli
  - Università Federico II, Cattedra di Oncologia Medica, Napoli
  - Casa di Cura La Maddalena, Palermo
  - Ospedale Silvestrini, Perugia
  - Ospedale Santa Chiara, Pisa
  - Università di Sassari, Sassari
  - Ospedale Santa Chiara, Trento
  - ASL Viterbo Ospedale Belcolle, Viterbo

REFERENCES:
- [Result] Rossi E, Morabito A, Di Rella F, Esposito G, Gravina A, Labonia V, Landi G, Nuzzo F, Pacilio C, De Maio E, Di Maio M, Piccirillo MC, De Feo G, D'Aiuto G, Botti G, Chiodini P, Gallo C, Perrone F, de Matteis A. Endocrine effects of adjuvant letrozole compared with tamoxifen in hormone-responsive postmenopausal patients with early breast cancer: the HOBOE trial. J Clin Oncol. 2009 Jul 1;27(19):3192-7. doi: 10.1200/JCO.2008.18.6213. Epub 2009 Apr 20. PMID 19380451
- [Result] Rossi E, Morabito A, De Maio E, Di Rella F, Esposito G, Gravina A, Labonia V, Landi G, Nuzzo F, Pacilio C, Piccirillo MC, D'Aiuto G, D'Aiuto M, Rinaldo M, Botti G, Gallo C, Perrone F, de Matteis A. Endocrine effects of adjuvant letrozole + triptorelin compared with tamoxifen + triptorelin in premenopausal patients with early breast cancer. J Clin Oncol. 2008 Jan 10;26(2):264-70. doi: 10.1200/JCO.2007.13.5319. Epub 2007 Dec 17. PMID 18086795
- [Result] Nuzzo F, Gallo C, Lastoria S, Di Maio M, Piccirillo MC, Gravina A, Landi G, Rossi E, Pacilio C, Labonia V, Di Rella F, Bartiromo A, Buonfanti G, De Feo G, Esposito G, D'Aniello R, Maiolino P, Signoriello S, De Maio E, Tinessa V, Colantuoni G, De Laurentiis M, D'Aiuto M, Di Bonito M, Botti G, Giordano P, Daniele G, Morabito A, Normanno N, de Matteis A, Perrone F. Bone effect of adjuvant tamoxifen, letrozole or letrozole plus zoledronic acid in early-stage breast cancer: the randomized phase 3 HOBOE study. Ann Oncol. 2012 Aug;23(8):2027-2033. doi: 10.1093/annonc/mdr600. Epub 2012 Mar 12. PMID 22412041
- [Derived] Gravina A, Gargiulo P, De Laurentiis M, Arenare L, De Placido S, Orditura M, Cinieri S, Riccardi F, Ribecco AS, Putzu C, Del Mastro L, Rossi E, Ciardiello F, Di Rella F, Nuzzo F, Pacilio C, Caputo R, Cianniello D, Forestieri V, Giuliano M, Arpino G, Orlando L, Mocerino C, Schettino C, Piccirillo MC, Gallo C, Perrone F. Ten-year update of HOBOE phase III trial comparing triptorelin plus either tamoxifen or letrozole or zoledronic acid + letrozole in premenopausal hormone receptor-positive early breast cancer patients. ESMO Open. 2025 Jan;10(1):104085. doi: 10.1016/j.esmoop.2024.104085. Epub 2025 Jan 3. PMID 39754976
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716
- [Derived] Perrone F, De Laurentiis M, De Placido S, Orditura M, Cinieri S, Riccardi F, Ribecco AS, Putzu C, Del Mastro L, Rossi E, Tinessa V, Mosconi AM, Nuzzo F, Di Rella F, Gravina A, Iodice G, Landi G, Pacilio C, Forestieri V, Lauria R, Fabbri A, Ibrahim T, De Maio E, Barni S, Gori S, Simeon V, Arenare L, Daniele G, Piccirillo MC, Normanno N, de Matteis A, Gallo C. Adjuvant zoledronic acid and letrozole plus ovarian function suppression in premenopausal breast cancer: HOBOE phase 3 randomised trial. Eur J Cancer. 2019 Sep;118:178-186. doi: 10.1016/j.ejca.2019.05.004. Epub 2019 Jun 1. PMID 31164265